CLINICAL TRIAL: NCT00000119
Title: Safety and Efficacy of a Heparin-Coated Intraocular Lens in Uveitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-15
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-09

CONDITIONS: Cataract; Uveitis
MeSH Terms: conditions — Cataract; Uveitis

INTERVENTIONS:
Device: Heparin Surface-Modified Intraocular Lens

SUMMARY:
To investigate the safety and efficacy of a heparin surface-modified intraocular lens in patients with uveitis undergoing cataract surgery.

To evaluate the safety and efficacy of intraocular lens implantation in patients with severe uveitis.

DETAILED DESCRIPTION:
Patients with uveitis are at high risk for significant complications following cataract surgery with intraocular lens implantation. Complications may result from the surgery itself or may develop after surgery as a result of the intraocular lens. Complications related to intraocular lens implantation include iris adhesions to the intraocular lens, which can result in lens capture; cellular deposits on the surface of the lens that can obscure vision; and uveitis. Recent studies have identified giant cells on the anterior surface of intraocular lenses in some patients with uveitis, appearing to indicate an intraocular lens-induced inflammatory response. Some of these patients have required multiple YAG laser procedures to remove these deposits.

Modification of the surface of the intraocular lens with a layer of heparin may provide a more biocompatible surface. Preclinical studies have shown a reduction in the degree of postoperative complications with the heparin surface-modified intraocular lens compared with an unmodified lens. Although retrospective case series have examined the use of heparin surface-modified intraocular lenses in patients with uveitis, a randomized, controlled clinical trial has not been performed.

This is a randomized clinical trial examining the safety and efficacy of the heparin surface-modified intraocular lens in patients with uveitis. Eighty patients with a history of uveitis in an eye requiring cataract surgery will be randomized to receive a heparin surface-modified intraocular lens or the same model of intraocular lens without surface modification. The primary end point of the study will be the development of cellular deposits on the anterior surface of the intraocular lens 1 year after surgery. These cellular deposits will be assessed by a masked grader using standard photographs. Secondary end points will include visual acuity, intraocular inflammation, development of anterior and posterior synechiae, and corneal endothelial cell counts.

ELIGIBILITY:
Women and men 18 years or older with a documented history of uveitis in an eye requiring cataract surgery are eligible for the study. In all patients, the eye must be free of active inflammation for at least 3 months before surgery, with or without anti-inflammatory medications. Exclusion criteria include corneal pathology or hazy media that preclude evaluation of the intraocular lens, uncontrolled glaucoma, and diabetes mellitus. Monocular patients and patients who cannot be followed for at least 1 year are also excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1994-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health, Bethesda, Maryland, United States